CLINICAL TRIAL: NCT03551691
Title: Proton Pump Inhibitors (PPI) and Fat Absorption in Subjects With Cystic Fibrosis (CF) and Exocrine Pancreatic Insufficiency (EPI)
Brief Title: Proton Pump Inhibitors (PPI) and Fat Absorption in Cystic Fibrosis (CF) and Exocrine Pancreatic Insufficiency (EPI)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: Chiesi USA, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 17-014666
Record Dates: First submitted 2018-05-29; First posted 2018-06-11 (Actual); Results first posted 2024-04-30 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: Pancreatic Insufficiency; Cystic Fibrosis
Keywords: fat absorption; pancreatic enzyme
MeSH Terms: conditions — Exocrine Pancreatic Insufficiency; Cystic Fibrosis | interventions — Omeprazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Omeprazole (Active Comparator): Subjects will take omeprazole 20mg daily for 28 days, then undergo assessments of fat absorption.
  Interventions: Drug: Omeprazole 20mg Capsule
- Placebo (Placebo Comparator): Subjects will take a placebo daily for 28 days, then undergo assessments of fat absorption.
  Interventions: Drug: Placebo oral capsule

INTERVENTIONS:
Drug: Omeprazole 20mg Capsule — Omeprazole 20mg daily for 28 days
  Other Names: PPI
  Arms: Omeprazole
Drug: Placebo oral capsule — Identically-appearing capsule to omeprazole for 28 days
  Other Names: Placebo
  Arms: Placebo

SUMMARY:
This is a clinical trial with a cross over design investigating the effect of the proton pump inhibitor omeprazole on fat malabsorption in subjects with cystic fibrosis and pancreatic insufficiency. Participants will be randomized to receive either omeprazole or placebo for 28 days, then cross over and receive omeprazole or placebo for another 28 days. Markers of fat absorption will be measured after each treatment course.

DETAILED DESCRIPTION:
Fat malabsorption contributes to poor nutritional status in people with cystic fibrosis (CF) and exocrine pancreatic insufficiency (EPI). Prescribing gastric acid-reducing agents such as proton pump inhibitors (PPIs) and histamine receptor antagonists (H2RAs) as an adjunct to pancreatic enzyme replacement therapy (PERT) to improve PERT efficacy and dietary fat absorption has become accepted clinical practice in CF, despite limited evidence to support the practice. Establishing the efficacy and true health benefit of acid suppression for nutritional status and outcomes in CF is particularly important in light of potential health risks and cost associated with long-term or even lifetime use of these medications.

This study aims to characterize changes in fat malabsorption using the coefficient of fat absorption (CFA) as the primary endpoint in subjects who are on and off acid suppression with a PPI in addition to PERT. Additionally, the SmartPill® will be used to evaluate duodenal power of hydrogen (pH) while on and off acid suppression, and the malabsorption blood test (MBT) will be used to characterize changes in fat absorption. Associations will be explored between changes in nutritional status (weight, height, BMI), clinical GI symptoms, and quality of life in subjects treated with PPI vs. placebo.

ELIGIBILITY:
Inclusion Criteria:

* Cystic fibrosis and pancreatic insufficiency (Fecal elastase <200 ug/g stool)
* Age ≥12 years
* In usual state of good health
* Willing to participate in a four-month study with three visits

Exclusion Criteria:

* Forced expiratory vital capacity at one second (FEV1) <40% predicted
* Pregnancy or breast feeding
* Other illness affecting growth or nutritional status
* Unwillingness to continue their clinically established PERT dose for the duration of the study
* Use of other medication that affects dietary fat absorption
* Allergy to soy products
* Allergy to safflower products
* For subjects ≥18 years, celiac disease or allergy to gluten

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2018-08-07 (Actual); Primary Completion 2022-11-02 (Actual); Study Completion 2022-11-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Virginia A Stallings, MD, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported will be shared upon request, after deidentification.
Supporting Information: Study Protocol, ICF
Time Frame: The data will be available immediately upon publication.
Access Criteria: Contact brownellj@email.chop.edu. Requestors will need to sign a data access agreement.

REFERENCES:
- [Background] Borowitz DS, Grand RJ, Durie PR. Use of pancreatic enzyme supplements for patients with cystic fibrosis in the context of fibrosing colonopathy. Consensus Committee. J Pediatr. 1995 Nov;127(5):681-4. doi: 10.1016/s0022-3476(95)70153-2. No abstract available. PMID 7472816
- [Background] Ng SM, Moore HS. Drug therapies for reducing gastric acidity in people with cystic fibrosis. Cochrane Database Syst Rev. 2016 Aug 22;2016(8):CD003424. doi: 10.1002/14651858.CD003424.pub4. PMID 27546383
- [Background] Stallings VA, Mondick JT, Schall JI, Barrett JS, Wilson M, Mascarenhas MR. Diagnosing malabsorption with systemic lipid profiling: pharmacokinetics of pentadecanoic acid and triheptadecanoic acid following oral administration in healthy subjects and subjects with cystic fibrosis. Int J Clin Pharmacol Ther. 2013 Apr;51(4):263-73. doi: 10.5414/CP201793. PMID 23357842
- [Background] Mascarenhas MR, Mondick J, Barrett JS, Wilson M, Stallings VA, Schall JI. Malabsorption blood test: Assessing fat absorption in patients with cystic fibrosis and pancreatic insufficiency. J Clin Pharmacol. 2015 Aug;55(8):854-65. doi: 10.1002/jcph.484. Epub 2015 Mar 23. PMID 25689042
- [Background] Lightdale JR, Gremse DA; Section on Gastroenterology, Hepatology, and Nutrition. Gastroesophageal reflux: management guidance for the pediatrician. Pediatrics. 2013 May;131(5):e1684-95. doi: 10.1542/peds.2013-0421. Epub 2013 Apr 29. PMID 23629618
- [Background] Heijerman HG, Lamers CB, Bakker W, Dijkman JH. Improvement of fecal fat excretion after addition of omeprazole to pancrease in cystic fibrosis is related to residual exocrine function of the pancreas. Dig Dis Sci. 1993 Jan;38(1):1-6. doi: 10.1007/BF01296765. PMID 8420740
- [Background] Heijerman HG, Lamers CB, Bakker W. Omeprazole enhances the efficacy of pancreatin (pancrease) in cystic fibrosis. Ann Intern Med. 1991 Feb 1;114(3):200-1. doi: 10.7326/0003-4819-114-3-200. PMID 1984743
- [Background] Proesmans M, De Boeck K. Omeprazole, a proton pump inhibitor, improves residual steatorrhoea in cystic fibrosis patients treated with high dose pancreatic enzymes. Eur J Pediatr. 2003 Nov;162(11):760-3. doi: 10.1007/s00431-003-1309-5. Epub 2003 Sep 17. PMID 13680386
- [Background] Cox KL, Isenberg JN, Osher AB, Dooley RR. The effect of cimetidine on maldigestion in cystic fibrosis. J Pediatr. 1979 Mar;94(3):488-92. doi: 10.1016/s0022-3476(79)80609-5. PMID 423042
- [Background] Carroccio A, Pardo F, Montalto G, Iapichino L, Soresi M, Averna MR, Iacono G, Notarbartolo A. Use of famotidine in severe exocrine pancreatic insufficiency with persistent maldigestion on enzymatic replacement therapy. A long-term study in cystic fibrosis. Dig Dis Sci. 1992 Sep;37(9):1441-6. doi: 10.1007/BF01296016. PMID 1505293
- [Background] Boyle BJ, Long WB, Balistreri WF, Widzer SJ, Huang N. Effect of cimetidine and pancreatic enzymes on serum and fecal bile acids and fat absorption in cystic fibrosis. Gastroenterology. 1980 May;78(5 Pt 1):950-3. PMID 7380201
- [Background] Chalmers DM, Brown RC, Miller MG, Clarke PC, Kelleher J, Littlewood JM, Losowsky MS. The influence of long-term cimetidine as an adjuvant to pancreatic enzyme therapy in cystic fibrosis. Acta Paediatr Scand. 1985 Jan;74(1):114-7. doi: 10.1111/j.1651-2227.1985.tb10930.x. PMID 3885675
- [Background] Bowler IM, Green JH, Wolfe SP, Littlewood JM. Resting energy expenditure and substrate oxidation rates in cystic fibrosis. Arch Dis Child. 1993 Jun;68(6):754-9. doi: 10.1136/adc.68.6.754. PMID 8333766
- [Background] Francisco MP, Wagner MH, Sherman JM, Theriaque D, Bowser E, Novak DA. Ranitidine and omeprazole as adjuvant therapy to pancrelipase to improve fat absorption in patients with cystic fibrosis. J Pediatr Gastroenterol Nutr. 2002 Jul;35(1):79-83. doi: 10.1097/00005176-200207000-00017. PMID 12142815
- [Background] Ng SM, Franchini AJ. Drug therapies for reducing gastric acidity in people with cystic fibrosis. Cochrane Database Syst Rev. 2014 Jul 13;(7):CD003424. doi: 10.1002/14651858.CD003424.pub3. PMID 25019293
- [Background] Ng SM, Francini AJ. Drug therapies for reducing gastric acidity in people with cystic fibrosis. Cochrane Database Syst Rev. 2012 Apr 18;(4):CD003424. doi: 10.1002/14651858.CD003424.pub2. PMID 22513912
- [Background] Ng SM, Jones AP. Drug therapies for reducing gastric acidity in people with cystic fibrosis. Cochrane Database Syst Rev. 2003;(2):CD003424. doi: 10.1002/14651858.CD003424. PMID 12804466
- [Background] Kaunitz JD, Akiba Y. Wireless telemetry and cystic fibrosis: just the pHacts. Dig Dis Sci. 2013 Aug;58(8):2129-30. doi: 10.1007/s10620-013-2714-x. Epub 2013 Jun 9. No abstract available. PMID 23748712
- [Background] Gelfond D, Ma C, Semler J, Borowitz D. Intestinal pH and gastrointestinal transit profiles in cystic fibrosis patients measured by wireless motility capsule. Dig Dis Sci. 2013 Aug;58(8):2275-81. doi: 10.1007/s10620-012-2209-1. Epub 2012 May 17. PMID 22592630
- [Background] Borowitz D, Baker SS, Duffy L, Baker RD, Fitzpatrick L, Gyamfi J, Jarembek K. Use of fecal elastase-1 to classify pancreatic status in patients with cystic fibrosis. J Pediatr. 2004 Sep;145(3):322-6. doi: 10.1016/j.jpeds.2004.04.049. PMID 15343184
- [Background] Borowitz D, Lin R, Baker SS. Comparison of monoclonal and polyclonal ELISAs for fecal elastase in patients with cystic fibrosis and pancreatic insufficiency. J Pediatr Gastroenterol Nutr. 2007 Feb;44(2):219-23. doi: 10.1097/MPG.0b013e31802c41de. PMID 17255835

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This is a randomized, cross-over study for which 19 participants were consented/enrolled; not all participants initiated study drug/placebo. Participants were randomized to receive placebo or drug first.
Pre-assignment Details: 19 subjects were randomized. There were 13 evaluable subjects who completed data collection at the end of the treatment period and 6 subjects did not complete data collection.
Groups:
- Study Drug First, Then Placebo: Subjects will take omeprazole 20mg daily for 28 days, then undergo assessments of fat absorption.
  Omeprazole 20mg Capsule: Omeprazole 20mg daily for 28 days
- Placebo First, Then Study Drug: Subjects will take a placebo daily for 28 days, then undergo assessments of fat absorption.
  Placebo oral capsule: Identically-appearing capsule to omeprazole for 28 days
Period: Overall Study
Arm/Group | Study Drug First, Then Placebo | Placebo First, Then Study Drug
Started | 9 | 10
Completed | 6 | 7
Not Completed | 3 | 3
Not completed — Withdrawal by Subject | 3 | 3

BASELINE CHARACTERISTICS:
Population: This randomized, crossover study includes baseline characteristics for 13 participants who both or either active and/or placebo treatment.
  Only data for 11 participants were available for analysis.
Groups:
- Total: Total of all reporting groups
Arm/Group | Study Drug First, Then Placebo | Placebo First, Then Study Drug | Total
Number analyzed (Participants) | 6 | 7 | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 19 (4) | 19 (4) | 19 (4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 7
  Male | 3 | 3 | 6
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White/Caucasian | 6 | 6 | 12
  African American | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Coefficient of Fat Absorption
Description: Gold standard measurement of fat malabsorption
Time Frame: After 28 days of treatment or placebo
Population: The primary outcome measurement (CFA) was not available for 2 participants who got study drug first and 2 participants who got placebo first.
Measure: Mean (Standard Deviation); unit: % fat absorption
Arm/Group | Omeprazole | Placebo
Number analyzed (Participants) | 7 | 4
% fat absorption | 80 (20) | 77 (16)

2. Secondary Outcome: Duodenal pH
Description: Change in duodenal pH as measured by the motility testing system (SmartPill)
Time Frame: After 28 days of treatment or placebo
Measure: Mean (Standard Deviation); unit: pH
Arm/Group | Omeprazole | Placebo
Number analyzed (Participants) | 4 | 4
pH | 6.03 (0.4) | 5.38 (0.8)

3. Secondary Outcome: Fat Absorption Via Malabsorption Blood Test
Description: Measurement of serum pentadecanoic acid and heptadecanoic acid
Time Frame: After 28 days of treatment or placebo
Measure: Mean (Standard Deviation); unit: mg*h/dl
Arm/Group | Omeprazole | Placebo
Number analyzed (Participants) | 9 | 9
mg*h/dl | 7.3 (2.1) | 9.6 (3.4)

ADVERSE EVENTS:
Time Frame: 28 days (while participant was on active treatment or placebo); total of 56 days.
Arm/Group | Omeprazole | Placebo
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/11
Other Adverse Events (participants affected / at risk) | 0/11 | 0/11

LIMITATIONS AND CAVEATS:
Analysis of the secondary measures remains ongoing and results are anticipated in the Spring of 2024. Results from secondary outcomes will be reported when data analysis are complete.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-12-11): https://cdn.clinicaltrials.gov/large-docs/91/NCT03551691/Prot_SAP_000.pdf